CLINICAL TRIAL: NCT01329341
Title: Service Dogs for Veterans With PTSD: A Randomized Clinical Trial
Brief Title: Service Dogs for Veterans With PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study concluded prematurly
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D8094-I
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: PTSD
Keywords: PTSD; Service Dogs
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Service Dogs
  Interventions: Other: Service Dogs

INTERVENTIONS:
Other: Service Dogs — Service dogs will be trained to help Veterans with PTSD

SUMMARY:
The purpose of this study is to evaluate use of service dogs for individuals who have been diagnosed with Post Traumatic Stress Disorder (PTSD). Objectives include: (1) assess the impact service dogs have on the mental health and quality of life of Veterans; (2) to provide recommendations to the VA to serve as guidance in providing service dogs to Veterans; and (3) To determine cost associated with total health care utilization and mental health care utilization among Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Referral from provider.
* PTSD diagnosis
* In active treatment for PTSD for at least three months at time of enrollment, with plans to remain in active treatment
* Acceptance by the dog vendor for the service dog
* Ability to adequately care for a dog - physically/financially
* Able to travel to vendor for pairing with dog

Exclusion Criteria:

* Been hospitalized for mental health reasons in the prior 6 months
* Not living at the same residence for 6 months.
* Diagnoses: Psychoses, Delusions, dementia, active alcohol/substance dependence. Moderate to severe TBI. Any other diagnosis deemed by PI to limit ability to participate or give informed consent
* At time of enrollment - Active suicidal ideation, homicide, cognitive disabilities that would preclude safety of animal and ability needed for participation in the study.
* Children under age 10 living in the home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie McGovern, RN, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Veterans were recruited prior to receipt of ServiceDog and given questionnaires to complete. They were followed and questionnaires completed every 3 months until receipt of Service Dog.
Period: Overall Study
Arm/Group | Arm 1
Started | 60
Completed | 16
Not Completed | 44
Not completed — Withdrawal by Subject | 44

BASELINE CHARACTERISTICS:
Groups:
- Service Dog: Veterans who received a service dog
Arm/Group | Service Dog
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 49
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Mental Health Outcomes
Description: Mental Health Outcomes are defined by the following measures: PCL-S - PTSD symptoms
Time Frame: 3,6,9,12,18 and 24 months after receipt of service dog
Population: No valid data to report.
Arm/Group | Service Dog
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from 7/1/2011 - 1/31/2017, 5 years, 7 months
Arm/Group | Service Dog
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 10/60
Other Adverse Events (participants affected / at risk) | 12/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Service Dog (N=60)
Subject death due to car accident (Injury, poisoning and procedural complications) | 1 (1) — Unknown what specific injuries caused the subject's death in the accident
Subject's child bitten by service dog (Skin and subcutaneous tissue disorders) | 1 (1) — Child had bruising, no medical attention required.
Subject paired with a service dog suffering from health problems. (Social circumstances) | 1 (1)
Subject fell down stairs at home and was hospitalized with a fractured ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Subject tripped over walker at home and sustained minor injuries - was treated at home by spouse (Skin and subcutaneous tissue disorders) | 1 (1) — skin tear and bruising occured
Subject twisted their ankle while on a walk and called 911. Was transported to the ER (Musculoskeletal and connective tissue disorders) | 1 (1) — Given medication and crutches in the ER and sent home
Subject hospitalized for removal of kidney related to cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Service dog euthanized due to inoperable spinal tumor (Social circumstances) | 1 (1)
Subject hospitalized (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject "not feeling right" and called 911. Hospitalized with respiratory difficulty. Monitored, treated and released after short inpatient stay.
Subject and service dog attacked by a dog (Skin and subcutaneous tissue disorders) | 1 (1) — Subject received minor puncture wound to finger and dog had injuries to his side. Both received outpatient medical treatment and released
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Service Dog (N=60)
Subject complaint about the veterinarian on the study team (Social circumstances) | 1 (1)
Subject divulged her phone number on a blog and received harassing calls (Social circumstances) | 1 (1)
Subject's child nipped by service dog (Social circumstances) | 1 (1) — No medical attention required
Subject's service dog died unexpectedly (Social circumstances) | 1 (1)
Subject's PHI sent to unsecure fax machine (Social circumstances) | 1 (1)
Financial exchange between subject and vendor (Social circumstances) | 1 (1) — Subject gave money to vendor to buy dog food and other items for dogs.
Vendor threatened subject with lawsuit over possession of puppy (Social circumstances) | 1 (1)
Vendor paired dog with subject prior to enrollement in study (Social circumstances) | 1 (1)
Subject's finger caught in service dog's leash and was injured (Musculoskeletal and connective tissue disorders) | 1 (1)
Subject upset that OIG was contacting him, felt harassed (Social circumstances) | 1 (1)
Veteran who withdrew from study upset about lack of insurance coverage (Social circumstances) | 1 (1)
Wife of subject shared withdrawal letter with others (Social circumstances) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated but a subsequent multisite clinical trial (NCT02039843) was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT01329341/Prot_SAP_000.pdf